CLINICAL TRIAL: NCT07152899
Title: New Approaches for the Treatment of Post-stroke Dysphagia and Dysphagia in Parkinson's Disease
Brief Title: Innovative Treatments for Neurogenic Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: ASST Santi Paolo e Carlo (Other); L. Sacco Department of Biomedical and Clinical Sciences, Milano, Italy (Unknown); Fondazione Don Carlo Gnocchi Onlus (Other); Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neu-Dysphagia
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-04

CONDITIONS: Stroke, Complication; Parkinson's Disease
Keywords: Dysphagia; Stroke; Parkinson's Disease; Transcranial Direct Current Stimulation (tDCS); Neuromuscular Electrical Stimulation (NMES); Swallowing Therapy
MeSH Terms: conditions — Stroke; Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Following informed consent, participants underwent a standardized evaluation protocol consisting of clinical and neurophysiological assessments. Swallowing function was assessed using the Dysphagia Outcome and Severity Scale (DOSS) as the primary outcome measure. Secondary outcomes include the Penetration-Aspiration Scale (PAS), Mann Assessment of Swallowing Ability (MASA), Swallowing Quality of Life Questionnaire (SWAL-QOL), and Motor Evoked Potentials (MEPs) of tongue musculature in a subgroup of participants.
  All stimulation interventions (tDCS or NMES) were delivered by trained clinicians according to standardized protocols. Each session was accompanied by a personalized intensive speech and swallowing therapy session, administered by certified speech-language pathologists.
Who Masked: Participant, Investigator
Masking Description: Participants, care providers, and outcome assessors will all be blinded to group allocation to ensure double-blind conditions throughout the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Unilateral anodal tDCS (Experimental): In post-stroke dysphagia
  Interventions: Other: Unilateral anodal tDCS
- Bihemispheric anodal tDCS (Experimental): In post-stroke dysphagia
  Interventions: Other: Bihemispheric anodal tDCS
- Sham tDCS (Placebo Comparator): In post-stroke dysphagia
  Interventions: Other: Sham tDCS
- Anodal tDCS in both hemispheres (Experimental): In Parkinson's disease dysphagia
  Interventions: Other: Bihemispheric anodal tDCS
- Placebo tDCS (Placebo Comparator): In Parkinson's disease dysphagia
  Interventions: Other: Sham tDCS
- NMES + swallowing therapy (Experimental): In patients with post-stroke dysphagia and Parkinson's disease dysphagia
  Interventions: Other: NMES + swallowing therapy
- Sham NMES + swallowing therapy (Placebo Comparator): In patients with post-stroke dysphagia and Parkinson's disease dysphagia
  Interventions: Other: Sham NMES + swallowing therapy

INTERVENTIONS:
Other: Unilateral anodal tDCS — Evaluates the effects of unilateral, anodal tDCS applied to the swallowing motor cortex in post-stroke patients with dysphagia
  Arms: Unilateral anodal tDCS
Other: Bihemispheric anodal tDCS — Evaluates the effects of bihemispheric, anodal tDCS applied to the swallowing motor cortex in post-stroke patients with dysphagia and in Parkinson's disease-related dysphagia
  Arms: Anodal tDCS in both hemispheres; Bihemispheric anodal tDCS
Other: Sham tDCS — Evaluates the effects of Sham tDCS applied to the swallowing motor cortex in post-stroke patients with dysphagia and in Parkinson's disease-related dysphagia
  Arms: Placebo tDCS; Sham tDCS
Other: NMES + swallowing therapy — Examines the effects of NMES therapy on swallowing function in both post-stroke and Parkinson's disease patients
  Arms: NMES + swallowing therapy
Other: Sham NMES + swallowing therapy — Examines the effects of Sham therapy on swallowing function in both post-stroke and Parkinson's disease patients
  Arms: Sham NMES + swallowing therapy

SUMMARY:
This study aims to evaluate different non-invasive and neuromuscular stimulation treatments for neurogenic dysphagia in post-stroke and Parkinson's disease patients. The study is divided into three sub-studies:

1. Unilateral, bihemispheric, or sham transcranial Direct Current Stimulation (tDCS) in post-stroke dysphagia (patients ≥2 weeks from onset).
2. Bihemispheric or sham tDCS in Parkinson's disease-related dysphagia.
3. Neuromuscular stimulation therapy in post-stroke and Parkinson's disease dysphagia.

DETAILED DESCRIPTION:
Neurogenic dysphagia, commonly seen in post-stroke and Parkinson's disease patients, significantly impacts quality of life. Despite emerging treatments, there remains a lack of consensus on the best approaches for these conditions. This study evaluates three different innovative therapeutic interventions and their efficacy in improving swallowing function:

Sub-study 1: Evaluates the effects of unilateral, bihemispheric, or sham tDCS applied to the swallowing motor cortex in post-stroke patients with dysphagia.

Sub-study 2: Evaluates the effects of bihemispheric or sham tDCS in Parkinson's disease patients with dysphagia.

Sub-study 3: Examines the effects of neuromuscular electrical stimulation (NMES) therapy on swallowing function in both post-stroke and Parkinson's disease patients.

Each intervention was administered over a 6-week period with outcome measures assessed at baseline and post-treatment. All treatments were applied in conjunction with a personalized and intensive speech therapy program.

This study aims to provide valuable insights into the effectiveness of tDCS and NMES as adjuncts to traditional swallowing therapy. By targeting mechanisms of brain plasticity and neuromuscular function, the study could improve treatment strategies for neurogenic dysphagia in stroke and Parkinson's disease patients. Ultimately, the findings could contribute to evidence-based guidelines for managing dysphagia in these populations.

This interventional study recruited a total of 110 participants: 70 patients with post-stroke dysphagia and 40 patients with Parkinson's disease-related dysphagia. Participants were consecutively enrolled from collaborating institutions.

Following informed consent, participants underwent a standardized evaluation protocol consisting of clinical and neurophysiological assessments. Swallowing function was assessed using the Dysphagia Outcome and Severity Scale (DOSS) as the primary outcome measure. Secondary outcomes include the Penetration-Aspiration Scale (PAS), Mann Assessment of Swallowing Ability (MASA), Swallowing Quality of Life Questionnaire (SWAL-QOL), and Motor Evoked Potentials (MEPs) of tongue musculature in a subgroup of participants.

All stimulation interventions (tDCS or NMES) were delivered by trained clinicians according to standardized protocols. Each session was accompanied by a personalized intensive speech and swallowing therapy session, administered by certified speech-language pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 years
* Diagnosis of post-stroke or Parkinson's disease-related dysphagia
* Dysphagia duration ≥ 2 weeks for post-stroke patients and ≥ 6 months for Parkinson's disease patients
* Ability to undergo rehabilitation therapy
* Written informed consent obtained

Exclusion Criteria:

* Severe dysphagia requiring Percutaneous Endoscopic Gastrostomy (PEG) feeding for more than 1 year
* Non-neurogenic causes of dysphagia
* Contraindications to tDCS or NMES
* Cognitive impairment affecting compliance with treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Dysphagia Outcome and Severity Scale (DOSS) score | At baseline and 6 weeks post-treatment
  Improvement in DOSS.The DOSS is a simple, easy-to-use, 7-point scale developed to systematically rate the functional severity of dysphagia based on objective assessment and make recommendations for diet level, independence level, and type of nutrition.

SECONDARY OUTCOMES:
Penetration-Aspiration Scale (PAS) score | At baseline and 6 weeks post-treatment
  Changes in PAS. It's a 8-point scale to score the degree of airway invasion and patient response.
Mann Assessment of Swallowing Ability (MASA) score | At baseline and 6 weeks post-treatment
  Clinical evaluation using the MASA. The MASA is an instrument that was designed for bedside evaluations for patients referred for swallowing function assessment.
  This assessment measures 24 different areas to gauge a patient's swallowing ability, in order to make appropriate recommendations for diet and fluid intake.
Swallowing Quality of Life (SWAL-QOL) questionnaire | At baseline and 6 weeks post-treatment
  The SWAL-QOL questionnaire was constructed for use in clinical research for patients with oropharyngeal dysphagia.
Motor Evoked Potentials (MEP) assessment | At baseline and 6 weeks post-treatment
  Motor Evoked Potentials (MEP) assessment of tongue muscle response in a small patients subgroup .

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cosentino, MD, Principal Investigator — Translational Neurophysiology
Locations (1):
- Translational Neurophysiology, Pavia, Italy

REFERENCES:
- [Background] Ahn YH, Sohn HJ, Park JS, Ahn TG, Shin YB, Park M, Ko SH, Shin YI. Effect of bihemispheric anodal transcranial direct current stimulation for dysphagia in chronic stroke patients: A randomized clinical trial. J Rehabil Med. 2017 Jan 19;49(1):30-35. doi: 10.2340/16501977-2170. PMID 27904911
- [Background] Arnold M, Liesirova K, Broeg-Morvay A, Meisterernst J, Schlager M, Mono ML, El-Koussy M, Kagi G, Jung S, Sarikaya H. Dysphagia in Acute Stroke: Incidence, Burden and Impact on Clinical Outcome. PLoS One. 2016 Feb 10;11(2):e0148424. doi: 10.1371/journal.pone.0148424. eCollection 2016. PMID 26863627
- [Background] Frost J, Robinson HF, Hibberd J. A comparison of neuromuscular electrical stimulation and traditional therapy, versus traditional therapy in patients with longstanding dysphagia. Curr Opin Otolaryngol Head Neck Surg. 2018 Jun;26(3):167-173. doi: 10.1097/MOO.0000000000000454. PMID 29553959
- [Background] Geeganage C, Beavan J, Ellender S, Bath PM. Interventions for dysphagia and nutritional support in acute and subacute stroke. Cochrane Database Syst Rev. 2012 Oct 17;10:CD000323. doi: 10.1002/14651858.CD000323.pub2. PMID 23076886
- [Background] Ginocchio D, Alfonsi E, Mozzanica F, Accornero AR, Bergonzoni A, Chiarello G, De Luca N, Farneti D, Marilia S, Calcagno P, Turroni V, Schindler A. Cross-Cultural Adaptation and Validation of the Italian Version of SWAL-QOL. Dysphagia. 2016 Oct;31(5):626-34. doi: 10.1007/s00455-016-9720-z. Epub 2016 Jul 21. PMID 27444734
- [Background] O'Neil KH, Purdy M, Falk J, Gallo L. The Dysphagia Outcome and Severity Scale. Dysphagia. 1999 Summer;14(3):139-45. doi: 10.1007/PL00009595. PMID 10341109
- [Background] Kumar S, Wagner CW, Frayne C, Zhu L, Selim M, Feng W, Schlaug G. Noninvasive brain stimulation may improve stroke-related dysphagia: a pilot study. Stroke. 2011 Apr;42(4):1035-40. doi: 10.1161/STROKEAHA.110.602128. Epub 2011 Mar 24. PMID 21441148
- [Background] Langmore SE, Pisegna JM. Efficacy of exercises to rehabilitate dysphagia: A critique of the literature. Int J Speech Lang Pathol. 2015 Jun;17(3):222-9. doi: 10.3109/17549507.2015.1024171. Epub 2015 Mar 31. PMID 25825989
- [Background] Liang Y, Lin J, Wang H, Li S, Chen F, Chen L, Li L. Evaluating the Efficacy of VitalStim Electrical Stimulation Combined with Swallowing Function Training for Treating Dysphagia following an Acute Stroke. Clinics (Sao Paulo). 2021 Nov 8;76:e3069. doi: 10.6061/clinics/2021/e3069. eCollection 2021. PMID 34755758
- [Background] Mann G, Hankey GJ, Cameron D. Swallowing function after stroke: prognosis and prognostic factors at 6 months. Stroke. 1999 Apr;30(4):744-8. doi: 10.1161/01.str.30.4.744. PMID 10187872
- [Background] Robbins J, Butler SG, Daniels SK, Diez Gross R, Langmore S, Lazarus CL, Martin-Harris B, McCabe D, Musson N, Rosenbek J. Swallowing and dysphagia rehabilitation: translating principles of neural plasticity into clinically oriented evidence. J Speech Lang Hear Res. 2008 Feb;51(1):S276-300. doi: 10.1044/1092-4388(2008/021). PMID 18230851
- [Background] Shigematsu T, Fujishima I, Ohno K. Transcranial direct current stimulation improves swallowing function in stroke patients. Neurorehabil Neural Repair. 2013 May;27(4):363-9. doi: 10.1177/1545968312474116. Epub 2013 Feb 7. PMID 23392916
- [Background] Speyer R, Baijens L, Heijnen M, Zwijnenberg I. Effects of therapy in oropharyngeal dysphagia by speech and language therapists: a systematic review. Dysphagia. 2010 Mar;25(1):40-65. doi: 10.1007/s00455-009-9239-7. Epub 2009 Sep 17. PMID 19760458
- [Background] Suntrup-Krueger S, Ringmaier C, Muhle P, Wollbrink A, Kemmling A, Hanning U, Claus I, Warnecke T, Teismann I, Pantev C, Dziewas R. Randomized trial of transcranial direct current stimulation for poststroke dysphagia. Ann Neurol. 2018 Feb;83(2):328-340. doi: 10.1002/ana.25151. Epub 2018 Feb 6. PMID 29350775
- [Background] Yang EJ, Baek SR, Shin J, Lim JY, Jang HJ, Kim YK, Paik NJ. Effects of transcranial direct current stimulation (tDCS) on post-stroke dysphagia. Restor Neurol Neurosci. 2012;30(4):303-11. doi: 10.3233/RNN-2012-110213. PMID 22572022